CLINICAL TRIAL: NCT06292234
Title: External Distraction Using Patient Specific Implant Versus Miniplates for Advancement of Hypoplastic Maxilla in Non-growing Cleft Patients
Brief Title: Patient Specific Implant Versus Miniplates for Advancement of Hypoplastic Maxilla
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar Mahmoud Ahmed Mohamed, Principal investigator, Phd candidate, Department of Oral & Maxillofacial Surgery, Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OMFS
Record Dates: First submitted 2024-02-25; First posted 2024-03-05 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Cleft Lip and Palate
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Intervention Model Description: Parallel randomized controlled trial with 1:1 allocation ratio and superiority framework
Who Masked: Participant
Masking Description: single blinded clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient specific implants (Experimental): Custom made designed implants
  Interventions: Device: PSI
- miniplates (Active Comparator): Over the counter miniplates
  Interventions: Device: Conventional miniplates

INTERVENTIONS:
Device: PSI — Fabrication of PSI implants using virtual surgical planning
  Arms: patient specific implants
Device: Conventional miniplates — Ready made miniplates
  Arms: miniplates

SUMMARY:
Distraction osteogenesis is the treatment of choice in management of severe maxillary anteroposterior deficiency allowing for a progressive bone generation and simultaneous expansion of the surrounding scarred soft tissue & better long-term stability & less relapse rate.

DETAILED DESCRIPTION:
Maxillary distraction using rigid external distraction device (RED) with skeletal anchorage in cleft lip and palate overcomes the disadvantages of tooth brone RED & showed reliable advancement & reasonable relapse rate in the short & long-term follow up & most importantly it solved somehow counterclockwise rotation of maxilla but still it can occur. Positioning of plates in relation to center of resistance of maxilla to adjust vector of distraction can be done now by using Virtual surgical planning (VSP) & fabrication of patient specific implants (PSI) to overcome problems encountered with use of conventional miniplates during distraction process. Limited data in literature with no randomized clinical trials were done to assess distraction effectiveness using PSI in RED with skeletal anchorage and its effect on velopharyngeal insufficiency (VPI) & speech. Based on that data, the research will compare distraction effectiveness, VPI & speech between using either PSI implants or miniplates for distraction.

ELIGIBILITY:
Inclusion Criteria:

1. Non growing cleft patients, age range (18-30 years)
2. Unilateral or bilateral cleft patients
3. Anteroposterior deficiency (1.5-2.5 cm)
4. No sex predilection

Exclusion Criteria:

1. Syndromic patients.
2. bone metabolism & systemic diseases.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Distraction effectiveness | immediate postoperative, 4 months postoperatively, 10 months postoperatively
  Amount of distraction using Lateral Cephalometry & FBCT measured in millimeters (mm)

SECONDARY OUTCOMES:
Velopharyngeal insufficiency | Preoperative , 4 months postoperatively, 10 months postoperatively
  Scoring from 0 to 4; 0: Normal, 1: minimal, 2: mild, 3: moderate, 4: sever using endoscopy
Speech | preoperative, 4 months postoperatively, and 10 months postoperatively
  Nasometry Speech assessment; 1=absent, 2=mild, 3=mild to moderate, 4=moderate, 5=moderate to severe and 6=severe.
Operative time | Immediate postoperative
  Measuring the time of the procedures in minutes
Wound dehiscence | immediate postoperative till 4 months postoperatively
  Clinical assessment of presence or absence of wound dehiscence (Binary: Yes or No)
Infection | immediate postoperative till 4 months postoperatively
  Clinical assessment of presence or absence of infection (Binary: Yes or No)
Nerve affection | immediate postoperative till 4 months postoperatively
  Clinical assessment of presence or absence of nerve affection (Binary: Yes or No)
Screw loosening | immediate postoperative till 4 months postoperatively
  Clinical assessment of presence or absence of screw loosening (Binary: Yes or No)
Overall complications | immediate postoperative, 4 months postoperatively and 10 months postoperatively
  Clinical assessment of presence or absence of complications (Binary: Yes or No)

IPD SHARING:
Plan to Share IPD: No